CLINICAL TRIAL: NCT04522414
Title: PremCry Study : Study of Ontogeny of Crying in Preterm Infants.
Acronym: PremCry
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN212020
Record Dates: First submitted 2020-08-03; First posted 2020-08-21 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Preterm Birth
Keywords: Newborn; ontogeny of crying; preterm infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infant
  Interventions: Other: cries longitudinally registered

INTERVENTIONS:
Other: cries longitudinally registered — Their cries will be longitudinally registered from the age of birth to the return home using an automatic record device: Song Meter SM4.

SUMMARY:
Crying is a survival mechanism for babies and their almost exclusive means of expression until the age of 4 months. Babies 'cry is mostly related to pain, a feeling of hunger, discomfort or separation following the departure of a parent around. Crying is a complex but essential means of communication and information between a baby and his parents that raises the question of their meaning.

Very few longitudinal studies have been produced on preterm's crying. As the term approaches, the characteristics of preterm babies' crying are similar to those of term infants. But these studies date back more than 30 years and are obsolete in terms of the quality and performance of sound recording equipment and signal processing.

No study has looked at the genesis of the cry itself and the varieties of the cry of the preterm baby, depending on whether it was in a situation of hunger, pain, discomfort (bath).

DETAILED DESCRIPTION:
This longitudinal study recordings of crying babies from 26 amenorrhea week to 33 amenorrhea week, 24 hours per week, each week until the return home. In the same time, parents will be asked to know the situation of the baby (hunger, pain, bath).

ELIGIBILITY:
Inclusion Criteria:

* Infant born between 26 and 33 amenorrhea week
* Live infant at birth
* Parent affiliated or entitled to a social security scheme
* Parent who received informed written information about the study

Exclusion Criteria:

- Intubated infant

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant born between 26 and 33 amenorrhea week will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Analysis fundamental frequency (f0) | at the end of hospitalization (on average 2 months)
  Measured by PRAAT software for 24h every week

SECONDARY OUTCOMES:
Analysis roughness of the cry (PC1) | at the end of hospitalization (on average 2 months)
  Measured by PRAAT software for 24h every week
Analysis pitch of the cry (PC2) | at the end of hospitalization (on average 2 months)
  Measured by PRAAT software for 24h every week
Analysis NIP∑ (neonatal index of parasympathetic activity) index | at the end of hospitalization (on average 2 months)
  Measured by monitor MDoloris® for 24h every week
Correlation between crying acoustic structures and parent's responses | at the end of hospitalization (on average 2 months)
  Measured by completed questionnaire by parents (Linear Mixed Model) every week

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No